CLINICAL TRIAL: NCT02109926
Title: A Multicentric Case-control Study to Assess the Association Between Environmental, Domestic and Occupational Exposures During Antenatal and Early Postnatal Periods and the Risk to Develop a Testicular Germ Cell Tumor During Adulthood
Brief Title: A Case-control Study to Assess the Association Between Environmental, Domestic and Occupational Exposures and the Risk of Testicular Germ Cell Tumor
Acronym: TESTIS
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TESTIS; ET14-004 (Other: Sponsor's number); 140184B-12 (Other: ANSM's number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Testicular Germ Cell Tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma and buffy coat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cases: testicular cancer patients
  Interventions: Other: Phone interview and blood test
- Group A controls: Sperm donors and husbands of women with fertility disorders All controls must have a normal spermogram
  Interventions: Other: Phone interview and blood test
- Group B controls: Husbands of women with a pathological pregnancy
  Interventions: Other: Phone interview and blood test

INTERVENTIONS:
Other: Phone interview and blood test — Subjects will be interviewed about environmental, domestic and occupational exposures during several periods of life Two blood samples will be collected at enrollment to study genetic polymorphisms

SUMMARY:
The incidence of testicular germ cell tumors, the most common cancer in men aged 15 to 45 years, has doubled in France in 30 years. Reasons remain unclear but a role of environmental factors, especially during critical periods of development, is strongly suspected. Reliable data on environmental exposure during this critical period are sparse.The discordant findings and the limitations of available studies underline the importance to conduct studies with sufficient statistical power to detect risk due to exposures during critical windows of vulnerability.

We conduct a multicentric case-control study to assess this association. Cases and controls will be enrolled during a 18-month period. They will be interviewed by professional telephone interviewers about their occupational and residential history and about their domestic exposure to pesticides and other nuisances.

An optional biological study to assess genetic polymorphisms known to be associated with testicular cancer will be proposed to every cases and controls.

Mothers (or close relative) of cases and controls will also be contacted (with son's agreement). If they agree to participate, they will also be interviewed about antenatal and early life exposure of their sons to pesticides and other nuisances.

Cases will be matched up with 2 controls (one of each group) both on age (+/- 2 years) and on recruiting center.

DETAILED DESCRIPTION:
Environmental exposure to pesticides will be assessed from subject's residential history, using a Geographic Information System.

Occupational exposure to pesticides and other nuisances will be assessed by an industrial hygienist who will be in charge to encode all subjects and mothers' occupations.

Domestic exposure to pesticides will be assessed from type, target and frequency of domestic pesticide use.

Based on these 3 sources of exposure, a score of exposition will be calculated for each case and each control.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 44 years old
* Born in metropolitan France
* Able to understand, read and write French
* Without any psychiatric and severe cognitive disorder
* Willingness to participate to the study
* Who has signed and dated an inform consent form
* Affiliated to a health care system

Exclusion Criteria:

* Who has a legal guardian
* History of testicular germ cell tumor or cryptorchidism (only for controls)

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases are patients with a testicular germ cell tumor. They will be recruited in the French infertility centers at the moment of sperm cryopreservation.
  Group A controls are sperm donors and husbands of women with fertility troubles. They will be recruited in the French infertility centers and in the medically assisted procreation centers.
  Group B controls are husbands of women followed for a pathological pregnancy. This group of controls will be recruited in the level III maternities.
Sampling Method: Non-Probability Sample
Enrollment: 1367 (Actual)
Dates: Start 2015-01; Primary Completion 2018-03-30 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Assess the association between pesticide exposure during Antenatal and Early Postnatal Periods and the risk of testicular cancer during adulthood | at the end of enrollment (18 months)
  Occupational, environmental and domestic exposures to pesticides and other nuisances will be assessed.

SECONDARY OUTCOMES:
Assess the association between a combined exposure to pesticides and the risk of testicular cancer during adulthood | at the end of enrollment (18 months)
  The association will be assessed during antenatal, postnatal early life and later life (adolescence and adulthood).
  Occupational, environmental and domestic exposures to pesticides and other nuisances will be assessed.
Analyse polymorphisms known to be associated with testicular cancer risk to explore gene-environment interactions | one year after the end of enrollment
  Polymorphisms involved in organochlorine metabolism pathways will also be assessed.
  Biological study

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice FERVERS, MD, Principal Investigator — Centre Leon Berard; Joachim SCHÜZ, PhD, Study Director — International Agency for Research on Cancer
Locations (22):
- France (22):
  - CHRU Jean Minjoz, Besançon
  - CHU Jean Verdier, Bondy
  - Maternité CHU Pellegrin, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - CHU de Caen, Caen
  - CHU Estaing, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU de Grenoble - Hôpital Couple Enfants, Grenoble
  - CHRU Lille - Hôpital Calmette, Lille
  - Centre Léon Bérard, Lyon
  - CHU La Conception, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Maternité Université Régionale, Nancy
  - CHU de Nice - Hôpital l'Archet, Nice
  - Hôpital Cochin, Paris
  - Hôpital Tenon, Paris
  - Hôpital Maison Blanche, Reims
  - CHU de Rennes - Hôpital Sud, Rennes
  - CHU Charles Nicolle, Rouen
  - Centre Médico-Chirurgical Obstétrique, Schiltigheim
  - Hôpital Paule de Viguier, Toulouse
  - CHU Bretonneau, Tours

REFERENCES:
- [Background] Belot A, Grosclaude P, Bossard N, Jougla E, Benhamou E, Delafosse P, Guizard AV, Molinie F, Danzon A, Bara S, Bouvier AM, Tretarre B, Binder-Foucard F, Colonna M, Daubisse L, Hedelin G, Launoy G, Le Stang N, Maynadie M, Monnereau A, Troussard X, Faivre J, Collignon A, Janoray I, Arveux P, Buemi A, Raverdy N, Schvartz C, Bovet M, Cherie-Challine L, Esteve J, Remontet L, Velten M. Cancer incidence and mortality in France over the period 1980-2005. Rev Epidemiol Sante Publique. 2008 Jun;56(3):159-175. doi: 10.1016/j.respe.2008.03.117. Epub 2008 Jun 10. PMID 18547762
- [Background] Bray F, Richiardi L, Ekbom A, Forman D, Pukkala E, Cuninkova M, Moller H. Do testicular seminoma and nonseminoma share the same etiology? Evidence from an age-period-cohort analysis of incidence trends in eight European countries. Cancer Epidemiol Biomarkers Prev. 2006 Apr;15(4):652-8. doi: 10.1158/1055-9965.EPI-05-0565. PMID 16614105
- [Background] Dalgaard MD, Weinhold N, Edsgard D, Silver JD, Pers TH, Nielsen JE, Jorgensen N, Juul A, Gerds TA, Giwercman A, Giwercman YL, Cohn-Cedermark G, Virtanen HE, Toppari J, Daugaard G, Jensen TS, Brunak S, Rajpert-De Meyts E, Skakkebaek NE, Leffers H, Gupta R. A genome-wide association study of men with symptoms of testicular dysgenesis syndrome and its network biology interpretation. J Med Genet. 2012 Jan;49(1):58-65. doi: 10.1136/jmedgenet-2011-100174. Epub 2011 Dec 3. PMID 22140272
- [Background] Kanetsky PA, Mitra N, Vardhanabhuti S, Li M, Vaughn DJ, Letrero R, Ciosek SL, Doody DR, Smith LM, Weaver J, Albano A, Chen C, Starr JR, Rader DJ, Godwin AK, Reilly MP, Hakonarson H, Schwartz SM, Nathanson KL. Common variation in KITLG and at 5q31.3 predisposes to testicular germ cell cancer. Nat Genet. 2009 Jul;41(7):811-5. doi: 10.1038/ng.393. Epub 2009 May 31. PMID 19483682
- [Background] Kratz CP, Han SS, Rosenberg PS, Berndt SI, Burdett L, Yeager M, Korde LA, Mai PL, Pfeiffer R, Greene MH. Variants in or near KITLG, BAK1, DMRT1, and TERT-CLPTM1L predispose to familial testicular germ cell tumour. J Med Genet. 2011 Jul;48(7):473-6. doi: 10.1136/jmedgenet-2011-100001. Epub 2011 May 26. PMID 21617256
- [Background] Rapley EA, Turnbull C, Al Olama AA, Dermitzakis ET, Linger R, Huddart RA, Renwick A, Hughes D, Hines S, Seal S, Morrison J, Nsengimana J, Deloukas P; UK Testicular Cancer Collaboration; Rahman N, Bishop DT, Easton DF, Stratton MR. A genome-wide association study of testicular germ cell tumor. Nat Genet. 2009 Jul;41(7):807-10. doi: 10.1038/ng.394. Epub 2009 May 31. PMID 19483681
- [Background] Turnbull C, Rapley EA, Seal S, Pernet D, Renwick A, Hughes D, Ricketts M, Linger R, Nsengimana J, Deloukas P, Huddart RA, Bishop DT, Easton DF, Stratton MR, Rahman N; UK Testicular Cancer Collaboration. Variants near DMRT1, TERT and ATF7IP are associated with testicular germ cell cancer. Nat Genet. 2010 Jul;42(7):604-7. doi: 10.1038/ng.607. Epub 2010 Jun 13. PMID 20543847
- [Background] Chia VM, Li Y, Quraishi SM, Graubard BI, Figueroa JD, Weber JP, Chanock SJ, Rubertone MV, Erickson RL, McGlynn KA. Effect modification of endocrine disruptors and testicular germ cell tumour risk by hormone-metabolizing genes. Int J Androl. 2010 Aug 1;33(4):588-96. doi: 10.1111/j.1365-2605.2009.00975.x. Epub 2009 Jul 20. PMID 19627379
- [Background] Garner MJ, Turner MC, Ghadirian P, Krewski D. Epidemiology of testicular cancer: an overview. Int J Cancer. 2005 Sep 1;116(3):331-9. doi: 10.1002/ijc.21032. PMID 15818625
- [Background] Pukkala E, Weiderpass E. Socio-economic differences in incidence rates of cancers of the male genital organs in Finland, 1971-95. Int J Cancer. 2002 Dec 20;102(6):643-8. doi: 10.1002/ijc.10749. PMID 12448008
- [Background] Swerdlow AJ, Skeet RG. Occupational associations of testicular cancer in south east England. Br J Ind Med. 1988 Apr;45(4):225-30. doi: 10.1136/oem.45.4.225. PMID 3377998
- [Background] Swerdlow AJ, Douglas AJ, Huttly SR, Smith PG. Cancer of the testis, socioeconomic status, and occupation. Br J Ind Med. 1991 Oct;48(10):670-4. doi: 10.1136/oem.48.10.670. PMID 1931725
- [Background] Van den Eeden SK, Weiss NS, Strader CH, Daling JR. Occupation and the occurrence of testicular cancer. Am J Ind Med. 1991;19(3):327-37. doi: 10.1002/ajim.4700190307. PMID 1848964
- [Background] Sarfati D, Shaw C, Blakely T, Atkinson J, Stanley J. Ethnic and socioeconomic trends in testicular cancer incidence in New Zealand. Int J Cancer. 2011 Apr 1;128(7):1683-91. doi: 10.1002/ijc.25486. Epub 2010 Jun 1. PMID 20518014
- [Background] Chia VM, Quraishi SM, Devesa SS, Purdue MP, Cook MB, McGlynn KA. International trends in the incidence of testicular cancer, 1973-2002. Cancer Epidemiol Biomarkers Prev. 2010 May;19(5):1151-9. doi: 10.1158/1055-9965.EPI-10-0031. PMID 20447912
- [Background] Doll R. Urban and rural factors in the aetiology of cancer. Int J Cancer. 1991 Apr 1;47(6):803-10. doi: 10.1002/ijc.2910470602. PMID 2010224
- [Background] Schouten LJ, Meijer H, Huveneers JA, Kiemeney LA. Urban-rural differences in cancer incidence in The Netherlands 1989-1991. Int J Epidemiol. 1996 Aug;25(4):729-36. doi: 10.1093/ije/25.4.729. PMID 8921449
- [Background] Sonneveld DJ, Schaapveld M, Sleijfer DT, Meerman GJ, van der Graaf WT, Sijmons RH, Koops HS, Hoekstra HJ. Geographic clustering of testicular cancer incidence in the northern part of The Netherlands. Br J Cancer. 1999 Dec;81(7):1262-7. doi: 10.1038/sj.bjc.6690839. PMID 10584892
- [Background] Walschaerts M, Muller A, Auger J, Bujan L, Guerin JF, Le Lannou D, Clavert A, Spira A, Jouannet P, Thonneau P. Environmental, occupational and familial risks for testicular cancer: a hospital-based case-control study. Int J Androl. 2007 Aug;30(4):222-9. doi: 10.1111/j.1365-2605.2007.00805.x. PMID 17708752
- [Background] Moller H. Work in agriculture, childhood residence, nitrate exposure, and testicular cancer risk: a case-control study in Denmark. Cancer Epidemiol Biomarkers Prev. 1997 Feb;6(2):141-4. PMID 9037566
- [Background] Rajpert-De Meyts E. Developmental model for the pathogenesis of testicular carcinoma in situ: genetic and environmental aspects. Hum Reprod Update. 2006 May-Jun;12(3):303-23. doi: 10.1093/humupd/dmk006. Epub 2006 Mar 15. PMID 16540528
- [Background] McGlynn KA, Trabert B. Adolescent and adult risk factors for testicular cancer. Nat Rev Urol. 2012 Apr 17;9(6):339-49. doi: 10.1038/nrurol.2012.61. PMID 22508459
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Main KM. Testicular dysgenesis syndrome: an increasingly common developmental disorder with environmental aspects. Hum Reprod. 2001 May;16(5):972-8. doi: 10.1093/humrep/16.5.972. PMID 11331648
- [Background] Akre O, Richiardi L. Does a testicular dysgenesis syndrome exist? Hum Reprod. 2009 Sep;24(9):2053-60. doi: 10.1093/humrep/dep174. Epub 2009 May 14. PMID 19443456
- [Background] Hemminki K, Li X. Cancer risks in Nordic immigrants and their offspring in Sweden. Eur J Cancer. 2002 Dec;38(18):2428-34. doi: 10.1016/s0959-8049(02)00496-3. PMID 12460788
- [Background] Myrup C, Westergaard T, Schnack T, Oudin A, Ritz C, Wohlfahrt J, Melbye M. Testicular cancer risk in first- and second-generation immigrants to Denmark. J Natl Cancer Inst. 2008 Jan 2;100(1):41-7. doi: 10.1093/jnci/djm276. Epub 2007 Dec 25. PMID 18159067
- [Background] Beranger R, Le Cornet C, Schuz J, Fervers B. Occupational and environmental exposures associated with testicular germ cell tumours: systematic review of prenatal and life-long exposures. PLoS One. 2013 Oct 14;8(10):e77130. doi: 10.1371/journal.pone.0077130. eCollection 2013. PMID 24155923
- [Background] Cohn BA, Cirillo PM, Christianson RE. Prenatal DDT exposure and testicular cancer: a nested case-control study. Arch Environ Occup Health. 2010 Jul-Sep;65(3):127-34. doi: 10.1080/19338241003730887. PMID 20705572
- [Background] Giannandrea F, Gandini L, Paoli D, Turci R, Figa-Talamanca I. Pesticide exposure and serum organochlorine residuals among testicular cancer patients and healthy controls. J Environ Sci Health B. 2011;46(8):780-7. doi: 10.1080/03601234.2012.597704. PMID 21902556
- [Background] Hardell L, Bavel B, Lindstrom G, Eriksson M, Carlberg M. In utero exposure to persistent organic pollutants in relation to testicular cancer risk. Int J Androl. 2006 Feb;29(1):228-34. doi: 10.1111/j.1365-2605.2005.00622.x. Epub 2005 Dec 20. PMID 16371110
- [Background] Kardaun JW, Hayes RB, Pottern LM, Brown LM, Hoover RN. Testicular cancer in young men and parental occupational exposure. Am J Ind Med. 1991;20(2):219-27. doi: 10.1002/ajim.4700200208. PMID 1951369
- [Background] Knight JA, Marrett LD. Parental occupational exposure and the risk of testicular cancer in Ontario. J Occup Environ Med. 1997 Apr;39(4):333-8. doi: 10.1097/00043764-199704000-00011. PMID 9113604
- [Background] Kristensen P, Andersen A, Irgens LM, Bye AS, Sundheim L. Cancer in offspring of parents engaged in agricultural activities in Norway: incidence and risk factors in the farm environment. Int J Cancer. 1996 Jan 3;65(1):39-50. doi: 10.1002/(SICI)1097-0215(19960103)65:13.0.CO;2-2. PMID 8543394
- [Background] Nori F, Carbone P, Giordano F, Osborn J, Figa-Talamanca I. Endocrine-disrupting chemicals and testicular cancer: a case-control study. Arch Environ Occup Health. 2006 Mar-Apr;61(2):87-95. doi: 10.3200/AEOH.61.2.87-95. PMID 17649960
- [Background] Rodvall Y, Dich J, Wiklund K. Cancer risk in offspring of male pesticide applicators in agriculture in Sweden. Occup Environ Med. 2003 Oct;60(10):798-801. doi: 10.1136/oem.60.10.798. PMID 14504372
- [Background] Provost D, Cantagrel A, Lebailly P, Jaffre A, Loyant V, Loiseau H, Vital A, Brochard P, Baldi I. Brain tumours and exposure to pesticides: a case-control study in southwestern France. Occup Environ Med. 2007 Aug;64(8):509-14. doi: 10.1136/oem.2006.028100. Epub 2007 May 30. PMID 17537748
- [Background] Chester G, Ward RJ. Occupational exposure and drift hazard during aerial application of paraquat to cotton. Arch Environ Contam Toxicol. 1984 Sep;13(5):551-63. doi: 10.1007/BF01056333. No abstract available. PMID 6486883
- [Background] Gunier RB, Ward MH, Airola M, Bell EM, Colt J, Nishioka M, Buffler PA, Reynolds P, Rull RP, Hertz A, Metayer C, Nuckols JR. Determinants of agricultural pesticide concentrations in carpet dust. Environ Health Perspect. 2011 Jul;119(7):970-6. doi: 10.1289/ehp.1002532. Epub 2011 Feb 17. PMID 21330232
- [Background] Koch D, Lu C, Fisker-Andersen J, Jolley L, Fenske RA. Temporal association of children's pesticide exposure and agricultural spraying: report of a longitudinal biological monitoring study. Environ Health Perspect. 2002 Aug;110(8):829-33. doi: 10.1289/ehp.02110829. PMID 12153767
- [Background] Ward MH, Lubin J, Giglierano J, Colt JS, Wolter C, Bekiroglu N, Camann D, Hartge P, Nuckols JR. Proximity to crops and residential exposure to agricultural herbicides in iowa. Environ Health Perspect. 2006 Jun;114(6):893-7. doi: 10.1289/ehp.8770. PMID 16759991
- [Background] Weppner S, Elgethun K, Lu C, Hebert V, Yost MG, Fenske RA. The Washington aerial spray drift study: children's exposure to methamidophos in an agricultural community following fixed-wing aircraft applications. J Expo Sci Environ Epidemiol. 2006 Sep;16(5):387-96. doi: 10.1038/sj.jea.7500461. Epub 2005 Oct 12. PMID 16249796
- [Background] Butte W, Heinzow B. Pollutants in house dust as indicators of indoor contamination. Rev Environ Contam Toxicol. 2002;175:1-46. PMID 12206053
- [Background] Zou B, Wilson JG, Zhan FB, Zeng Y. Air pollution exposure assessment methods utilized in epidemiological studies. J Environ Monit. 2009 Mar;11(3):475-90. doi: 10.1039/b813889c. Epub 2009 Feb 13. PMID 19280026
- [Derived] Guth M, Coste A, Lefevre M, Deygas F, Danjou A, Ahmadi S, Dananche B, Perol O, Boyle H, Schuz J, Bujan L, Metzler-Guillemain C, Giscard d'Estaing S, Teletin M, Ducrocq B, Frapsauce C, Olsson A, Charbotel B, Fervers B; TESTIS study group. Testicular germ cell tumour risk by occupation and industry: a French case-control study - TESTIS. Occup Environ Med. 2023 Jul;80(7):407-417. doi: 10.1136/oemed-2022-108601. Epub 2023 May 25. PMID 37230752